CLINICAL TRIAL: NCT04243980
Title: Short Term Results of Short Anatomical Femoral Stem in Total Hip Arthroplasty - Prospective Study
Brief Title: Anatomical Femoral Stem in Total Hip Arthroplasty
Acronym: THR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raja Hakim, Medical Doctor, HaEmek Medical Center, Israel
Other Study IDs: EMC-19-0100
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Patient Compliance; Patient Satisfaction
MeSH Terms: conditions — Patient Compliance; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients after total hip arthroplasty with short femoral stem
  Interventions: Device: Short anatomical femoral stem in THR

INTERVENTIONS:
Device: Short anatomical femoral stem in THR — Patients with osteoarthritis after total hip arthroplasty

SUMMARY:
A study that detect the femoral anteversion after total hip arthroplasty using short anatomical femoral stem compared to the contrast side

ELIGIBILITY:
Inclusion Criteria:

* age 18-90
* patients who had THR as an elective surgery
* patients who had THR with short femoral anatomical stem

Exclusion Criteria:

* severe osteoporosis with Dorr C classification
* s/p bilateral hip arthroplasty
* non-complaint patients
* revision surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged 18 - 90 who had THR as an elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Femoral anteversion | Post-Operatively, through study completion, an average of 2 years
  comparing femoral anteversion after THR using CT scan

SECONDARY OUTCOMES:
Harris Hip Score | 6 weeks, 3 month, 6 month post-operative
  The HHS is a physician-completed instrument that consists of subscales for pain severity (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 0-4 points), and range of motion (2 items, 0-5 points).
  Where a score < 70 indicating a poor result and those of 90-100 indicating an excellent result

IPD SHARING:
Plan to Share IPD: No